CLINICAL TRIAL: NCT05846490
Title: Impact of Obstructive Sleep Apnea Treatment on Blood Pressure Control in Chronic Kidney Disease: A Randomized Trial
Brief Title: Impact of Obstructive Sleep Apnea (OSA) Treatment on Blood Pressure Control in Chronic Kidney Disease
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Luciano F Drager, MD, PhD, Associate Professor of Medicine, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 64401922.8.0000.0068
Record Dates: First submitted 2023-04-14; First posted 2023-05-06 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Sleep Apnea; Chronic Kidney Diseases
MeSH Terms: conditions — Sleep Apnea Syndromes; Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Continuous positive airway pressure (CPAP) (Experimental): Standard OSA treatment + BP adjustments with anti-hypertensive therapy
  Interventions: Device: CPAP
- Usual Care (Active Comparator): BP adjustments with anti-hypertensive therapy
  Interventions: Drug: Usual care

INTERVENTIONS:
Device: CPAP — Continuous positive airway pressure + anti-hypertensive treatment intensification (if necessary)
  Arms: Continuous positive airway pressure (CPAP)
Drug: Usual care — Anti-hypertensive treatment intensification (if necessary)
  Arms: Usual Care

SUMMARY:
The role of obstructive sleep apnea (OSA) on chronic kidney disease (CKD) is not clear. This randomized clinical trial will test the impact of OSA treatment on blood pressure (BP) and on the estimated glomerular filtration rate (eGFR) in patients with CKD IIIb and IV (eGFR 44-15 ml/min). A polygraph will be performed to assess the presence of OSA (defined by an apnea-hypopnea index ≥15 events/hour). Patients with OSA will be randomized to use continuous positive upper airway pressure (CPAP) or to maintain optimized clinical treatment for BP control. Antihypertensive medication adjustments will be allowed using a standard protocol for both groups by the same researcher, who will not have access to CPAP follow-up. In addition to clinical (including BP and ambulatory BP monitoring, ABPM) and laboratory assessments at baseline, we will follow up at 3 months, 6 months, 9 months and 12 months after randomization of the proposed outcomes. Target organ damage analyses, such as the retina and echocardiography, will be performed at baseline and after 1 year of randomization. Primary objective: to compare the effect of CPAP on the need to adjust antihypertensive medication to control systolic BP (<130mmHg) in patients with CKD; secondary objectives: 1) to evaluate the reduction in systolic and diastolic BP by office and ABPM; 2) assessment of nocturnal BP dipping; 3) to evaluate the impact of OSA treatment with CPAP on eGFR during follow-up; 4) to evaluate the impact of OSA treatment with CPAP on the evolution of albuminuria; 5) assessment of other target organ damage such as retinopathy and cardiac remodeling; 6) to evaluate the impact of OSA treatment with CPAP on the possible delay for renal replacement therapy or end-stage renal disease (eGFR <15ml/min and dialysis); 7) to evaluate the impact of OSA treatment with CPAP on the quality of life of patients with CKD. With a significance level of 5% and study power of 90%, two-tailed hypothesis testing, 74 patients with OSA per group, i.e., 148 patients in total, will be required to assess the primary endpoint (we estimate that 25% and 50% of patients in control and CPAP groups will not need to adjust their antihypertensive medication at follow-up, respectively).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of hypertension: Use of oral antihypertensive drugs or systolic BP (SBP) >140 mmHg and/or diastolic BP (DBP) >90 mmHg on 2 office measurements or >130x80 mmHg (24 hours ABPM).
* eGFR by the CKD-EPI equation between 45 ml/min/1.73m2 and 15 ml/min/1.73m2 (in conservative treatment of CKD).

Exclusion Criteria:

* Professional drivers;
* Home supplemental oxygen users;
* Patients under current treatment for OSA;
* Pregnant women;
* Patients with malignant neoplasms or terminal illnesses;
* Severe asthma or chronic obstructive pulmonary disease;
* Patients with systemic lupus erythematosus, amyloidosis or systemic sclerosis;
* Patients with a history of solid organ transplants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Anti-hypertensive intensification | 1 year
  Percentage of patients that required treatment modification aiming at blood pressure control

SECONDARY OUTCOMES:
Systolic and diastolic blood pressure change by office measurement and ambulatory blood pressure monitoring | 1 year
  Absolute blood pressure change
Nocturnal blood pressure dipping | 1 year
  Assessment of nocturnal blood pressure dipping using ambulatory blood pressure monitoring
Estimated glomerular filtration rate (eGFR) | 1 year
  Impact of OSA treatment with CPAP on eGFR
Albuminuria | 1 year
  Impact of OSA treatment with CPAP on the evolution of albuminuria
Target organ damage using echocardiogram and fundoscopy | 1 year
  Impact of OSA treatment with CPAP on target organ damage such as grade of retinopathy and cardiac remodeling (left ventricular mass index, diastolic dysfunction, etc. by echocardiography).
End-stage renal disease (need of dialysis) | 1 year
  Impact of OSA treatment with CPAP on the possible delay for renal replacement therapy or end-stage renal disease (eGFR <15ml/min)
Continuous analysis of Quality of life | 1 year
  Impact of OSA treatment with CPAP on the quality of life (measured by 36-Item Short Form Health Survey). The lowest and highest possible scores are 0 and 100, respectively. The lower the score the higher impairment in quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Luciano Drager, MD, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Fernanda Trani Ferreira, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided